CLINICAL TRIAL: NCT02448745
Title: Liberia Insecticide Treated Durable Wall Linings Study: Protocol for a Cluster Randomised Trial (DL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Mentor Initiative (Other)
Collaborators: Ministry of Health, Liberia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LiberiaDL
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Malaria, Falciparum; Anemia
MeSH Terms: conditions — Malaria, Falciparum; Anemia

ARMS (2):
- Control (No Intervention): 21 clusters composed of one or more villages with a total number of 30 to 70 children under 5 years old. Routine distribution of long-lasting insecticidal nets is the only malaria control intervention.
- Intervention (Experimental): 21 clusters composed of one or more villages with a total of 30 to 70 children under 5 years old. Routine distribution of long-lasting insecticidal nets is available and in addition insecticide treated wall lining is installed in all sleeping areas with homeowner consent. All 4 walls and the ceiling are covered with lining.
  Interventions: Device: Insecticide treated wall lining

INTERVENTIONS:
Device: Insecticide treated wall lining — Polypropylene non-woven fabric.
  Other Names: Durable wall lining; PermaNet Lining
  Arms: Intervention

SUMMARY:
A cluster-randomized control trial will study the effect of insecticide-treated wall lining on malaria transmission in Bomi County, Liberia. Half of the villages enrolled in the study will receive insecticide-treated wall lining covering their walls and ceilings in addition to long-lasting insecticidal nets, while the other half will be protected by existing long-lasting insecticidal nets.

DETAILED DESCRIPTION:
Long-lasting insecticidal nets (LLINs) are the established vector control product for malaria control. In Bomi County Liberia, LLINs have been distributed but malaria prevalence in children under 5 remains high, with prevalence in study villages found to be 42% in April 2014. The major malaria vector species are resistant to pyrethroid insecticides approved for use in LLINs, and new control measures with non-pyrethroid active ingredients may protect the population.

ELIGIBILITY:
Inclusion Criteria:

* Child resides in village
* Child presents with parent or guardian

Exclusion Criteria:

* Child or guardian has history of Ebola exposure
* Child has 3 symptoms of Ebola

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6317 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Malaria Prevalence | 6 months
  Tested by mRDT and PCR

SECONDARY OUTCOMES:
Hemoglobin | 6 months
  Hemoglobin measured by Hemocue 301
Fever | 6 months
  Number of participants with Fever, defined as tympanic temperature above 37.5C
Mosquito biting rate. | 2 months
  Mosquitoes trapped indoors and outdoors using light traps and exit traps.

CONTACTS AND LOCATIONS:
Overall Officials: David J Giesbrecht, MSc, Principal Investigator — Study Coordinator
Locations (1):
- Bomi County Health Team, Tubmanburg, Bomi County, Liberia

REFERENCES:
- [Derived] Giesbrecht D, Belleh TG, Pontarollo J, Hinneh VS, Pratt O, Kamal S, Allan R. Durable wall lining for malaria control in Liberia: results of a cluster randomized trial. Malar J. 2023 Jan 12;22(1):15. doi: 10.1186/s12936-022-04429-7. PMID 36635660
- See also: The MENTOR Initiative — http://www.thementorinitiative.org/